CLINICAL TRIAL: NCT00631475
Title: Open-Label Extension Study in Patients With Idiopathic Pulmonary Fibrosis Who Completed Protocol AC-052-321 (NCT00391443)
Brief Title: Open Label Extension Study in Patients With Idiopathic Pulmonary Fibrosis Who Completed Protocol AC-052-321/ BUILD 3 / NCT00391443
Acronym: BUILD OL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-322
Record Dates: First submitted 2008-02-12; First posted 2008-03-07 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Actelion; Idiopathic Pulmonary Fibrosis; bosentan; Tracleer; Interstitial Lung Disease; BUILD 3 (NCT00391443)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): For patients who were administered bosentan during BUILD 3 (NCT00391443):
  Same dose will continue
  For patients who were administered placebo during BUILD 3 (NCT00391443):
  Initial dose: 62.5 mg for 4 weeks Maintenance dose: 125 mg
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — For patients who were administered Bosentan during BUILD 3 (NCT00391443):
  continue on same dose
  For patients who were administered placebo during BUILD 3 (NCT00391443):
  Oral Bosentan 62.5 mg for 4 weeks; maintenance dose: 125 mg ( 62.5 if patient weighs < 90 lbs.)
  Other Names: Tracleer

SUMMARY:
This Open-label extension study in patients with Idiopathic Pulmonary Fibrosis who completed protocol AC-052-321 / BUILD 3 (NCT00391443) will asses the long term safety and tolerability of bosentan in patients with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

Patients should have completed all the assessments from the BUILD 3 (NCT00391443) end of study (EOS) visit.

* Signed informed consent prior to initiation of any study-related procedures.
* Women of childbearing potential must have a negative serum pregnancy test and use reliable methods of contraception during study treatment and for 3 months after study treatment termination.

Exclusion Criteria:

* Any major violation of protocol AC-052-321 / BUILD 3 (NCT00391443).
* Pregnancy or breast-feeding.
* AST and/or ALT > 3 times the upper limit of the normal range.
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results, such as drug or alcohol dependence or psychiatric disease.
* Known hypersensitivity to bosentan or any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Leconte, Study Chair — Actelion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 61 centers in 15 countries (Australia, Belgium, Canada, Czech Republic, France, Germany, Ireland, Israel, Italy, Japan, South Korea, , Spain, Switzerland, UK, and USA. The first patient started on 5 March 2008 and the last patient, last visit was on 01 April 2010.
Pre-assignment Details: In total, 128 of the 615 patients who received randomized treatment in BUILD 3 (NCT00391443) rolled over into the BUILD 3 OL extension.
Groups:
- Bosentan Treatment: Oral bosentan 62.5 mg twice daily (b.i.d.) for the first 4 weeks, and oral bosentan 125 mg b.i.d. (62.5 mg b.i.d. if </= 40 kg) thereafter
Period: Overall Study
Arm/Group | Bosentan Treatment
Started | 128
Completed | 83
Not Completed | 45
Not completed — Death | 18
Not completed — Adverse Event | 14
Not completed — Withdrew consent | 5
Not completed — Preparation for lung transplant | 8

BASELINE CHARACTERISTICS:
Arm/Group | Bosentan Treatment
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.2)
Age, Customized [Number; unit: participants]
  18-40 years | 1
  41-60 years | 33
  61-70 years | 62
  >70 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 97
Region of Enrollment [Number; unit: participants]
  Australia | 12
  Belgium | 1
  Canada | 14
  Czech Republic | 1
  France | 3
  Germany | 11
  Ireland | 1
  Israel | 4
  Italy | 2
  Japan | 8
  Korea, Republic of | 5
  Spain | 8
  Switzerland | 4
  United Kingdom | 3
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Extent of Exposure to Bosentan in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Description: Mean extent of exposure to bosentan treatment in months
Time Frame: Start of study to end of study, up to 21 months
Population: For two patients, the exact treatment stop date was missing and the duration could not be calculated, but these patients received at least 345 and 127 days of open label (OL) treatment.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bosentan Treatment
Number analyzed (Participants) | 126
months | 6.4 (4.6)

2. Secondary Outcome: Number of Patients Exposed to Bosentan Over Time
Description: Numbers of participants exposed to bosentan treatment over time
Time Frame: Start to end of study, up to 21 months
Population: For two patients, the exact treatment stop date was missing and the duration could not be calculated, but these patients received at least 345 and 127 days of OL treatment, respectively.
Measure: Number; unit: Participants
Arm/Group | Bosentan Treatment
Number analyzed (Participants) | 126
Participants
  For at least 4 months | 74
  For at least 8 months | 44
  For at least 12 months | 17
  For at least 16 months | 7
  For at least 20 months | 2

3. Secondary Outcome: Adverse Events (AE) Leading to Discontinuation of Study Drug.
Description: Number of participants with at least one AE that led to permanent discontinuation of study treatment.
Time Frame: Start to end of study, up to 21 months
Population: Study population
Measure: Number; unit: participants
Arm/Group | Bosentan Treatment
Number analyzed (Participants) | 128
participants | 32

4. Secondary Outcome: Treatment-emergent Serious Adverse Events (SAE)
Description: Number of participants with at least one SAE during the study.
Time Frame: up to 21 months plus 28 days after the end of study drug
Population: Study population
Measure: Number; unit: participants
Arm/Group | Bosentan Treatment
Number analyzed (Participants) | 128
participants | 51

5. Secondary Outcome: Occurrence of Liver Function Test (LFT: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)) Abnormality.
Description: Number of participants with an increase in ALT and/or AST to > 3 times upper limit of normal during the study.
Time Frame: up to 21 months, plus 24 hours after the end of study treatment
Population: Study population
Measure: Number; unit: participants
Arm/Group | Bosentan Treatment
Number analyzed (Participants) | 128
participants | 3

ADVERSE EVENTS:
Time Frame: Up to 28 days after the end of study drug
Description: Only adverse events leading to premature discontinuation of study treatment were reported during the study. All serious adverse events occurring during and up to 28 days after end-of-study treatment were reported. Events listed as idiopathic pulmonary fibrosis were reported as worsening of idiopathic pulmonary fibrosis.
Arm/Group | Bosentan Treatment
Serious Adverse Events (participants affected / at risk) | 51/128
Other Adverse Events (participants affected / at risk) | 5/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan Treatment (N=128)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 23
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Coronary artery disease (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Blood iron decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Lung transplant (Surgical and medical procedures) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Renal colic (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan Treatment (N=128)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Actelion, with steering committee, shall complete the review and provide any modifications required to protect Actelion's patent rights and confidential information within sixty (60) days of receipt of the proposed publication. During this period, Investigator shall not permit publication. If Actelion reasonably anticipates filing a patent application claiming an invention arising out of the Study, such publication shall be delayed until after the application is filed.